CLINICAL TRIAL: NCT02028546
Title: The Effect of Bathing and Moisturizers on Skin Hydration in Atopic Dermatitis: an in Vivo Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Srinakharinwirot University (Other)
Responsible Party: Principal Investigator, Arisa Kaewkes, Doctor, Srinakharinwirot University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Srinakharinwirot fund
Record Dates: First submitted 2013-12-19; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis, skin cleansing, cleanser, moisturizer, skin hydration
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Baths

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Water (Experimental): The patients in water group were soaking an arm for 10 minutes with tap water before application of moisturizer. (Excepted the 4th regimen included no bathing, waited for 10 minutes and followed by moisturizer application.)
  Interventions: Procedure: bathing and moisturizer application
- mild cleanser (Experimental): The patients in mild cleanser group were soaking an arm for 10 minutes with mild cleanser before application of moisturizer. (Excepted the 4th regimen included no bathing, waited for 10 minutes and followed by moisturizer application.) Non soap base cleanser contained Sodium Cocoyl Isethionate was used in this mild cleanser arm.
  Interventions: Procedure: bathing and moisturizer application

INTERVENTIONS:
Procedure: bathing and moisturizer application — regimen 1: soaking an arm for 10 minutes, no moisturizer application regimen 2: soaking an arm for 10 minutes,immediate moisturizer application regimen 3: soaking an arm for 10 minutes, delayed moisturizer application for 30 min.
  regimen 4: wait for 10 minutes,no soaking, moisturizer application (moisturizer alone) (All regimens were completed in all patients with 2 visits (7 days interval))

SUMMARY:
The purpose of this study is to determine the hydration effect of various regimens of skin bathing and moisturizer application on atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* male or female;
* Age range 18-45 years;
* Subjects have history and physical findings consistent with mild to moderate AD with SCORAD score ≤ 40;
* Stop using some drugs such as oral corticosteroid for at least 4 weeks, topical corticosteroid and calcineurin inhibitor for at least 2 weeks, food supplement such as evening primrose oil, wheat extract Flax seed oil sunflowerseed oil, borage oil and fish oil for at least 3 months;
* Subjects who have signed the written informed consent.

Exclusion Criteria:

* Subjects who have medical histories such as zinc or essential fatty acid deficiency, end stage renal disease, hypothyroidism, human immunodeficiency virus (HIV), malignancies, obstructive biliary disease, diabetes mellitus and in those who have had radiation or other medical histories that may interfere the outcome;
* Subjects who ingest drugs that could interfere with the study results such as diuretics, antiandrogens, lipid reducing agents, isotretinoin cimetidine;
* Subjects cannot enroll until the end of the project;
* Subjects who have allergy to any ingredient in the moisturizer or cleanser that will be used in the protocol;
* Pregnant woman or lactating woman.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Skin hydration (skin capacitance) by using Corneometer and the trans-epidermal water loss value by using Tewameter of various regimens of bathing and moisturizer application | The skin hydration (capacitance value) and transepidermal water loss value were assessed at baseline and every 30 minutes for 120 minutes after each regimen.

SECONDARY OUTCOMES:
skin hydration (capacitance value) by using Corneometer and transepidermal water loss value by using Tewameter between immediate and delayed (30 minutes) moisturizer application after bathing. | The skin hydration (capacitance value) and TEWL value were assessed at baseline and every 30 minutes for 120 minutes after each regimen.

OTHER OUTCOMES:
Skin hydration(capacitance value) by using Corneometer and transepidermal water loss value by using Tewameter between water and mild cleanser | The skin hydration (capacitance value) and TEWL value were assessed at baseline and every 30 minutes for 120 minutes after each regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Arisa Kaewkes, MSc dermatology, Principal Investigator — Skin center, Faculty of Medicine, Srinakharinwirot University
Locations (1):
- Skin Center, Faculty of Medicine, Srinkharinwirot University, Bangkok, Bangkok, Thailand